CLINICAL TRIAL: NCT06484309
Title: The Effect of Reflexology on Perceived Perineal Pain During Episiotomy Repair.
Brief Title: Nonpharmacological Method for Relief During Episiotomy Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sena Dilek Aksoy, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: sdilek9
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pain
Keywords: Episiotomy; Reflexology; vaginal birth
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reflexology Group (Experimental): * Participants will sign an informed voluntary consent form during the active phase of labor,
  * Group assignment will be made,
  * Participant Information Form will be filled in,
  * The study will continue if episiotomy is performed at birth; If episiotomy is not performed at birth, it will not be included in the study.
  * Episiotomy repair will be performed by CG after anesthesia (5 ml lidocaine 2%) is applied in the 3rd stage of labor,
  * Reflexology application will be performed during episiotomy repair,
  * Evaluation with VAS will be performed before repair, during perineal repair (internal), during skin repair and immediately after the repair is completed,
  * The McGill Pain Questionnaire will be completed 20 minutes after episiotomy repair.
  Interventions: Behavioral: Reflexology Group
- Control group (No Intervention): * Participants will sign an informed voluntary consent form during the active phase of labor,
  * Group assignment will be made,
  * Participant Information Form will be filled in,
  * The study will continue if episiotomy is performed at birth; If episiotomy is not performed at birth, it will not be included in the study.
  * Episiotomy repair will be performed by CG after anesthesia (5 ml lidocaine 2%) is applied in the 3rd stage of labor,
  * Evaluation with VAS will be performed before repair, during perineal repair (internal), during skin repair and immediately after the repair is completed,
  * The McGill Pain Questionnaire will be completed 20 minutes after episiotomy repair.

INTERVENTIONS:
Behavioral: Reflexology Group — * In the 3rd stage of labor, local anesthesia (5 ml lidocaine 2%) will be applied and episiotomy repair will begin.
  * Reflexology application will be started at the same time,
  * Reflexology application will continue for at least 20-30 minutes during the episiotomy repair until the episiotomy repair is completed,
  * Pain will be evaluated with VAS to determine the pain level four times in total: just before suturing, during perineal suturing (internal), during skin suturing and immediately after suturing is completed,
  * Approximately 15-20 minutes after the end of the episiotomy repair, a face-to-face interview will be held and the McGill Pain Questionnaire will be filled out.
  Arms: Reflexology Group

SUMMARY:
The study was planned as a randomized controlled trial to evaluate the effect of reflexology on perceived perineal pain during episiotomy repair. The research will be carried out with participants who gave birth vaginally at Darıca Farabi Training and Research Hospital between July and December 2024. The research will be carried out with two groups: reflexology and control groups. Considering the sample size in the R pwrss (Statistical Power and Sample Size Calculation Tools) program, a type 1 (alpha) error of 0.05 and a power of 0.80, it was calculated that the study group should be at least 32 in the reflexology group and 32 in the control group. Considering the confounding variables, it was planned to recruit 25% more participants for each group, and therefore it was decided to recruit 40 participants per group. The participants included in the study will be divided into two groups by determining which group they will be included in from the website called "Random List", a random number generation program. Thus, each participant's number and group number will be determined and recorded. Research data will be collected using the Participant Information Form, VAS (Visual Analog Scale) and McGill Ağrı survey, which were created by the researcher within the framework of the literature on the subject. The data of the research will be evaluated using SPSS (IBM) 29.0 program. In evaluating the data; Descriptive statistics and comparative statistical analyzes will be used. Statistical significance level will be accepted as p<0.05.

DETAILED DESCRIPTION:
Aim: To examine the effect of reflexology on perceived perineal pain during episiotomy repair.

Hypothesis(s):

H0: There is no difference between the perineal pain of the group in which reflexology was applied and the group in which reflexology was not applied during episiotomy repair.

H1: There is a difference between the perineal pain of the group in which reflexology was applied and the group in which reflexology was not applied during episiotomy repair.

Type of Research: This study was designed as a randomized controlled experimental study.

In order to determine the sample size in the study, it was calculated according to the research conducted by Sharifi et al (2022). Considering the sample size in the R pwrss (Statistical Power and Sample Size Calculation Tools) program, a type 1 (alpha) error of 0.05 and a power of 0.80, it was calculated that the study group should be at least 32 in the reflexology group and 32 in the control group. Considering the confounding variables, it was planned to recruit 25% more participants for each group, and therefore it was decided to recruit 40 participants per group, 80 participants in total.

The participants included in the study will be divided into two groups by determining which group they will be included in from the website called "Random List", a random number generation program. Thus, each participant's number and group number will be determined and recorded.

Research data will be collected using the Participant Information Form, VAS (Visual Analog Scale) and McGill Pain questionnaire to assess pain during episiotomy repair.

Participant Information Form It was prepared by the researcher within the framework of the literature. The form consists of a total of 14 questions that question women's socio-demographic and obstetrics-related information.

VAS for Evaluation Pain during Episiotomy Repair: The participant marks his or her own pain on a 10 cm ruler, which is marked as "no pain" at one end and the most severe pain at the other end. The participant is told that there are two endpoints and to mark any place between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement. The VAS is more sensitive than the simple descriptive scale.

McGill Short Form for Assessment of Pain Following Episiotomy Repair: The McGill Pain Questionnaire was developed by Melzack and Torgerson and is used to evaluate pain multidimensionally. There are 15 criteria by which pain is evaluated. 11 of these criteria are to evaluate the emotional dimension of pain, and 4 are to evaluate the perceptual dimension of pain. Assessment of pain was rated on an intensity scale from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe). In the first part of the scale, a total of three pain scores are obtained: sensory pain score, perceptual pain score and total pain score. Sensory pain score ranges from 0-33, perceptual pain score ranges from 0-12, and total pain score ranges from 0-45. An increase in the score indicates that the pain also increases. Second Part: In this part, there are five word groups ranging from "mild pain" to "unbearable pain" to determine the severity of the patient's pain. Third Part: In the third part of MAS-CF, the patient's current pain intensity was evaluated using a visual comparison scale.

Application of Research After obtaining the necessary ethics committee and institutional permissions to conduct the research, the institution will be visited and participants who gave birth normally with episiotomy and meet the inclusion criteria for the study will be interviewed. Data will be collected by the researcher in the hospital delivery room. Women will be informed about the research and the purpose of the research will be explained. Those who agree to participate in the research will be asked to read and sign the Informed Consent Form. Participants who meet the criteria will be divided into reflexology and control groups. The website called "https://www.randomlists.com/", a random number generation program, will be used to determine the selection process. Thus, each participant's number and group number will be determined and recorded. Episiotomy repairs will be performed by the same midwife. We were going to do another investigative reflexology application. Data collection forms will be filled out by an independent midwife who is not involved in the research. One of the researchers, SDA, has approved international training and certification in the ability to apply foot reflexology techniques based on standard protocol.

For the reflexology group, first a 4-minute general massage will be applied to each foot, then a 2-minute specific reflexology will be applied in the form of rotational pressures to each point of the pelvis, sacrum, uterus and solar plexus. The application will take approximately 20-30 minutes. These points were agreed upon by experts in reflexology as effective points in reducing pain and anxiety. The control group will receive only general massage on each foot for 4 minutes.

Statistical analysis will be performed using IBM SPSS Statistic 29.0 (IBM Corp., Armonk, NY, USA). Descriptive statistical methods (number, percentage, mean, standard deviation) will be used in the evaluation of socio-demographic data. When the data is found to be suitable for normal distribution, parametric tests (chi-square, T test, etc.) will be used to compare categorical variables, and when the data is not found to be suitable for normal distribution, non-parametric tests (Mann-Whitney U Test) will be used. Statistical significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write,
* Those who have sufficient mental health to fill out the survey form,
* Between the ages of 18-35,
* Primiparous,
* At term gestational age (37-42 weeks),
* Having spontaneous birth with medial lateral episiotomy,
* The baby is healthy (does not require intervention or treatment),
* Participants who volunteered to participate in the study.

Exclusion Criteria:

* Those with visual, hearing or perception impairments,
* Having obstetric complications,
* Those who are allergic to anesthetic drugs and latex,
* Those with vaginal anomalies and signs of infection,
* Those with lacerations other than episiotomy (anal sphincter injury or 3rd or 4th degree laceration),
* Having an episiotomy smaller than 2 cm and larger than 4 cm,
* If the newborn is unhealthy or stillborn,
* Having a newborn who needs oxygen support,
* Possible bleeding or bleeding,
* Participants requiring large amounts of anesthesia during episiotomy repair.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale to assess episiotomy pain | 5 minutes before episiotomy repair
  The participant marks his or her pain on a 10 cm ruler; On one end it says no pain, on the other end it says worst pain. The participant is told that there are two extreme points and to mark any place between these points that corresponds to the severity of the pain. The distance between the pain stop and the point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in measuring pain intensity. VAS is more sensitive than the simple descriptive scale.
Visual analog scale to assess episiotomy pain | 10 minutes after episiotomy repair begins
  The participant marks his or her pain on a 10 cm ruler; On one end it says no pain, on the other end it says worst pain. The participant is told that there are two extreme points and to mark any place between these points that corresponds to the severity of the pain. The distance between the pain stop and the point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in measuring pain intensity. VAS is more sensitive than the simple descriptive scale.
Visual analog scale to assess episiotomy pain | 20 minutes after episiotomy repair begins
  The participant marks his or her pain on a 10 cm ruler; On one end it says no pain, on the other end it says worst pain. The participant is told that there are two extreme points and to mark any place between these points that corresponds to the severity of the pain. The distance between the pain stop and the point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in measuring pain intensity. VAS is more sensitive than the simple descriptive scale.
Visual analog scale to assess episiotomy pain | 5 minutes after episiotomy repair is completed
  The participant marks his or her pain on a 10 cm ruler; On one end it says no pain, on the other end it says worst pain. The participant is told that there are two extreme points and to mark any place between these points that corresponds to the severity of the pain. The distance between the pain stop and the point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in measuring pain intensity. VAS is more sensitive than the simple descriptive scale.

SECONDARY OUTCOMES:
McGill Pain Questionnaire to assess episiotomy pain | 20 minutes after episiotomy repair is completed
  The McGill Pain Questionnaire consists of three parts. The first part contains 15 descriptive word groups containing the characteristics of pain. 11 of these evaluate the sensory dimension of pain, and 4 evaluate the perceptual dimension. These descriptive words were rated on an intensity scale from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = excessive). In the first part of the scale, a total of three pain scores are obtained: sensory pain score, perceptual pain score and total pain score. In the second part, there are five word groups ranging from "mild pain" to "unbearable pain" to determine the severity of pain. In the third part, pain intensity is evaluated using a visual comparison scale. An increase in the score indicates that the pain also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Cemile Gokce, Midwife, Study Chair — Darica Farabi Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Darica Farabi Training and Research Hospital, Kocaeli
  - Kocaeli University, Kocaeli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharifi N, Bahri N, Hadizadeh-Talasaz F, Azizi H, Nezami H, Tohidinik HR. A randomized clinical trial on the effect of foot reflexology performed in the fourth stage of labor on uterine afterpain. BMC Pregnancy Childbirth. 2022 Jan 21;22(1):57. doi: 10.1186/s12884-022-04376-w. PMID 35062899